CLINICAL TRIAL: NCT01669811
Title: A Multicentre, Randomised, Double-blind, Parallel-group, Comparative Study to Compare the Efficacy and Safety of D961H 20 mg Twice Daily Oral Administration and D961H 20 mg Once Daily Oral Administration in Patients With Refractory Reflux Esophagitis
Brief Title: Compare D961H 20 mg Bid and 20 mg qd in Patients With Refractory Reflux Esophagitis (Inflammation of Lower Esophagus)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D961UC00002
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Refractory Reflux Esophagitis
Keywords: Refractory Reflux Esophagitis,; Japanese,; Nexium,; twice daily,; oral administration
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- D961H 20mg twice daily (Experimental): Double-blinded
  Interventions: Drug: Esomeprazole (D961H) twice daily
- D961H 20mg once daily (Active Comparator): Double-blinded
  Interventions: Drug: Esomeprazole (D961H) once daily

INTERVENTIONS:
Drug: Esomeprazole (D961H) twice daily — One capsule of esomeprazole 20 mg (in the form of esomeprazole magnesium salt) will be administered in the morning and in the evening
  Arms: D961H 20mg twice daily
Drug: Esomeprazole (D961H) once daily — One capsule of esomeprazole 20 mg (in the form of esomeprazole magnesium salt) will be administered in the morning and one corresponding placebo capsule in the evening
  Arms: D961H 20mg once daily

SUMMARY:
This is a phase 3 multicentre, randomised, double-blind, parallel-group, comparative study to evaluate the efficacy of esomeprazole (D961H) 20 mg twice daily and esomeprazole (D961H) 20 mg once daily in patients (in the form of esomeprazole magnesium salt) with refractory reflux esophagitis after 8 weeks of standard Proton-pump inhibitor (PPI) therapy by assessment of presence/absence of inflammation (esophagitis) at Week 8 according to the Los Angeles (LA) classification

DETAILED DESCRIPTION:
A multicentre, randomised, double-blind, parallel-group, comparative study to compare the efficacy and safety of D961H 20 mg twice daily oral administration and D961H 20 mg once daily oral administration in patients with refractory reflux esophagitis

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Patients with RE classified into LA classification Grade A, B, C or D by Endoscopy despite of at least 8-week treatment using standard doses of PPIs.
3. Patients must fulfill at least one of the following criteria such as (i) RE with LA grade C/D at Endoscopy on visit 1 and/or history of RE with LA grade C/D, (ii) RE was diagnosed more than 1 year before visit 1.
4. Patients who are able to complete the Patient Diary

Exclusion Criteria:

1. Male or female aged less than 20 years at the time of informed consent.
2. Patients with current evidence of the gastrointestinal diseases/conditions such as esophageal stricture to interfere with the evaluation of the study etc
3. Gastric or duodenal ulcer verified by Endoscopy within 12 weeks before randomisation.
4. Previous esophageal, gastric or duodenal surgery except simple closure of perforated ulcer, simple endoscopic treatment with simple operation etc
5. Current or historical evidence (within 12 weeks prior to randomisation) of the diseases/conditions as judged to interfere with the evaluation of the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tore Lind, MSD, Study Director — AstraZeneca, Moelndal, Sweden; Lan Chen, Study Director — AstraZeneca, Osaka, Japan; Yoshikazu Kinoshita, PROFESSOR OF MEDICINE, Principal Investigator — Dept of Gastroenterology and Hepatology, Shimane, Japan
Locations (63):
- Japan (63):
  - Research Site, Abiko-shi
  - Research Site, Adachi-ku
  - Research Site, Annaka-shi
  - Research Site, Asahikawa-shi
  - Research Site, Asakura-shi
  - Research Site, Beppu-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fujiidera-shi
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Hamamatsu
  - Research Site, Hirakata-shi
  - Research Site, Hitachi-shi
  - Research Site, Ibara-shi
  - Research Site, Ichiki-Kushikino-shi
  - Research Site, Ishikari-shi
  - Research Site, Iwata-shi
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kamakura-shi
  - Research Site, Kanazawa
  - Research Site, Karatsu-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kirishima-shi
  - Research Site, Kita-ku
  - Research Site, Kobe
  - Research Site, Kochi
  - Research Site, Koga-shi
  - Research Site, Koriyama-shi
  - Research Site, Kumagaya-shi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Machida-shi
  - Research Site, Matsumoto-shi
  - Research Site, Meguro-ku
  - Research Site, Moriguchi-shi
  - Research Site, Nishinomiya-shi
  - Research Site, Ogori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Otawara-shi
  - Research Site, Ōita
  - Research Site, Ōta-ku
  - Research Site, Saga
  - Research Site, Saitama-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakushu
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shibuya-ku
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takasaki-shi
  - Research Site, Takatsuki-shi
  - Research Site, Toshima-ku
  - Research Site, Toyama
  - Research Site, Uji-shi
  - Research Site, Wakayama
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
  - Research Site, Yufu-shi

REFERENCES:
- See also: D961UC00002_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=712&filename=D961UC00002_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 25 August 2012. Last subject completed on 30 May 2014.
Pre-assignment Details: Out of 1398 enrolled subjects, 287 subjects were randomised and 1111 subjects were not randomised. The reasons of no randomisation were 'Eligibilty criteria not met' (1067 subjects), 'Subject decision' (37 subjects), 'Adverse event' (2 subjects) and other reasons (5 subjects).
Groups:
- D961H 20 mg BID: Hard capsule containing 22.3 mg of D961H as enteric coated pellets
- D961H 20 mg QD + Placebo: Hard capsule unidentifiable to D961H capsule 20 mg
Period: Overall Study
Arm/Group | D961H 20 mg BID | D961H 20 mg QD + Placebo
Started | 145 | 142
Completed | 142 | 131
Not Completed | 3 | 11
Not completed — Investigator decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 2 | 6
Not completed — Eligibility Criteria Not Fulfilled | 0 | 2

BASELINE CHARACTERISTICS:
Population: It was found that 2 patients in D961H 20 mg QD + Placebo group had no refractory RE after randomisation. Therefore, these two patients were excluded from the full analysis set, which was the primary analysis set of this study and was used for summaries of baseline characteristics and outcome measures.
Groups:
- D961H 20 mg BID: D961H 20 mg twice Daily
- D961H 20 mg QD + Placebo: D961H 20 mg once daily along with placebo
- Total: Total of all reporting groups
Arm/Group | D961H 20 mg BID | D961H 20 mg QD + Placebo | Total
Number analyzed (Participants) | 145 | 140 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (13.87) [32 to 90] | 61.7 (14.72) [24 to 91] | 63.2 (14.35) [24 to 91]
Age, Customized [Number; unit: Participants]
  <65 | 68 | 69 | 137
  >=65 | 77 | 71 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 76 | 70 | 146
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 145 | 140 | 285

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Healing of RE Who Were Graded "O" at Week 8 Out of Participants Who Were Graded "A" to "D" at Baseline According to Los Angeles Classification
Description: Percentage of participants with healing of reflux esophagitis (RE) who were graded "O" (No RE) at Week 8 out of participants who were graded "A" (least severe) to "D" (most severe) at baseline according to Los Angeles classification
Time Frame: 8 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who had at least one dose of investigational product
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- D961H 20mg Bid: D961H 20mg twice daily
- D961H 20mg QD + Placebo: D961H 20mg once daily along with placebo
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 145 | 140
Percentage of participants | 92.4 [86.9 to 95.7] | 68.6 [60.5 to 75.7]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on healing of refractory RE in comparison with D20 qd; Test type: Superiority or Other; p < 0.0001, Chi-squared — p-value is obtained using chi square method; 95% CI is obtained using Newcombe-Wilson score method without continuity correction; Difference in proportions = 23.8, 95% CI 2-sided [14.9 to 32.6]

2. Secondary Outcome: Percentage of Participants With Healing of RE Who Were Graded "O" at Week 4 Out of Participants Who Were Graded "A" to "D" at Baseline According to Los Angeles Classification
Description: Percentage of participants with healing of reflux esophagitis (RE) who were graded "O" (No RE) at Week 4 out of participants who were graded "A" (least severe) to "D" (most severe) at baseline according to Los Angeles classification
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 145 | 140
Percentage of participants | 81.4 [74.3 to 86.9] | 48.6 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on healing of refractory RE in comparison with D20 qd; Test type: Superiority or Other; p < 0.0001, Chi-squared — p-value is obtained using chi square method; 95% CI is obtained using Newcombe-Wilson score method without continuity correction; Difference in proportions = 32.8, 95% CI 2-sided [21.9 to 42.6]

3. Secondary Outcome: Cumulative Percentage of Participants Who Had Sustained Resolution of GERD Symptom -Heartburn at Week 4
Description: Cumulative percentage of participants who had sustained resolution (defined as at least 7-day consecutive symptom free) of gastroesophageal reflux disease (GERD) symptom -heartburn at Week 4 (on Day 29) based on the Kaplan-Meier method.
Time Frame: 4 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who took at least one dose of investigational product. However, out of these participants, only participants who had the GERD symptom -heartburn at baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 90 | 81
Percentage of participants | 81.1 [74.3 to 86.9] | 72.8 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on gastroesophageal reflux disease (GERD) symptoms in comparison with D20 qd; Test type: Superiority or Other; p = 0.1452, Log Rank; 95% CI of the hazard ratio is obtained using Cox proportional hazards model including a factor of treatment group; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.91 to 1.83]

4. Secondary Outcome: Cumulative Percentage of Participants Who Had Sustained Resolution of GERD Symptom -Acid Regurgitation at Week 4
Description: Cumulative percentage of participants who had sustained resolution (defined as at least 7-day consecutive symptom free) of gastroesophageal reflux disease (GERD) symptom -acid regurgitation at Week 4 (on Day 29) based on the Kaplan-Meier method.
Time Frame: 4 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who took at least one dose of investigational product. However, out of these participants, only participants who had the GERD symptom -acid regurgitation at baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 78 | 67
Percentage of participants | 73.1 [74.3 to 86.9] | 61.2 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on gastroesophageal reflux disease (GERD) symptoms in comparison with D20 qd; Test type: Superiority or Other; p = 0.0837, Log Rank; 95% CI of the hazard ratio is obtained using Cox proportional hazards model including a factor of treatment group; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.97 to 2.18]

5. Secondary Outcome: Cumulative Percentage of Participants Who Had Sustained Resolution of GERD Symptom -Abdominal Pain at Week 4
Description: Cumulative percentage of participants who had sustained resolution (defined as at least 7-day consecutive symptom free) of gastroesophageal reflux disease (GERD) symptom -abdominal pain at Week 4 (on Day 29) based on the Kaplan-Meier method.
Time Frame: 4 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who took at least one dose of investigational product. However, out of these participants, only participants who had the GERD symptom -abdominal pain at baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 47 | 44
Percentage of participants | 68.1 [74.3 to 86.9] | 59.1 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on gastroesophageal reflux disease (GERD) symptoms in comparison with D20 qd; Test type: Superiority or Other; p = 0.2678, Log Rank; 95% CI of the hazard ratio is obtained using Cox proportional hazards model including a factor of treatment group; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.80 to 2.26]

6. Secondary Outcome: Cumulative Percentage of Participants Who Had Sustained Resolution of GERD Symptom -Difficulty of Swallowing at Week 4
Description: Cumulative percentage of participants who had sustained resolution (defined as at least 7-day consecutive symptom free) of gastroesophageal reflux disease (GERD) symptom -difficulty of swallowing at Week 4 (on Day 29) based on the Kaplan-Meier method.
Time Frame: 4 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who took at least one dose of investigational product. However, out of these participants, only participants who had the GERD symptom -difficulty of swallowing at baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 28 | 27
Percentage of participants | 78.6 [74.3 to 86.9] | 74.1 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on gastroesophageal reflux disease (GERD) symptoms in comparison with D20 qd; Test type: Superiority or Other; p = 0.6389, Log Rank; 95% CI of the hazard ratio is obtained using Cox proportional hazards model including a factor of treatment group; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.62 to 2.12]

7. Secondary Outcome: Cumulative Percentage of Participants Who Had Sustained Resolution of GERD Symptom -Sleep Disturbance at Week 4
Description: Cumulative percentage of participants who had sustained resolution (defined as at least 7-day consecutive symptom free) of gastroesophageal reflux disease (GERD) symptom -sleep disturbance at Week 4 (on Day 29) based on the Kaplan-Meier method.
Time Frame: 4 Weeks
Population: Included all of the randomised participants who were definitely diagnosed to have refractory RE before the randomisation and who took at least one dose of investigational product. However, out of these participants, only participants who had the GERD symptom -sleep disturbance at baseline were included.
Measure: Number; unit: Percentage of participants
Arm/Group | D961H 20mg Bid | D961H 20mg QD + Placebo
Number analyzed (Participants) | 34 | 28
Percentage of participants | 91.2 [74.3 to 86.9] | 89.3 [40.4 to 56.8]
Statistical Analysis 1: Comparison: D961H 20mg Bid vs D961H 20mg QD + Placebo; To evaluate the efficacy of D20 bid on gastroesophageal reflux disease (GERD) symptoms in comparison with D20 qd; Test type: Superiority or Other; p = 0.4485, Log Rank; 95% CI of the hazard ratio is obtained using Cox proportional hazards model including a factor of treatment group; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.80 to 2.38]

ADVERSE EVENTS:
Arm/Group | D961H 20 mg BID | D961H 20 mg QD + Placebo
Serious Adverse Events (participants affected / at risk) | 1/145 | 3/142
Other Adverse Events (participants affected / at risk) | 8/145 | 9/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D961H 20 mg BID (N=145) | D961H 20 mg QD + Placebo (N=142)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parotid abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D961H 20 mg BID (N=145) | D961H 20 mg QD + Placebo (N=142)
Nasopharyngitis (Infections and infestations) | 8 (8) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study withiout AZ approval before this study was completed.